CLINICAL TRIAL: NCT05072847
Title: Introduction of the ADAPT System for Pertrochanteric Fractures in an Orthopedic Department
Brief Title: Introduction of the ADAPT System in an Orthopedic Department
Acronym: ADAPTintro
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Per Gundtoft, Principal Investigator, Consultant, PhD, Aarhus University Hospital
Other Study IDs: ADAPT_1
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Pertrochanteric Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADAPT: The ADAPT system by Striker

SUMMARY:
The ADAPT system by Stryker is introduced in the orthopedic department (at Aarhus University Hospital). Following the introduction of the ADAPT system all pertrochanteric fractures operated with a gamma3 nail by stryker are operated with the use of the ADAPT system. Following surgery the operating surgeon fill out a questionaire on the use of ADAPT.

DETAILED DESCRIPTION:
At the ortopedic department, Aarhus University Hospital pertrochanteric fractures are mostly operated with the gamma3 system by Stryker.

The ADAPT system is software based instrumentation designed for use in Gamma3 surgery. The software assists the surgeon with implant alignment, lag screw length determination, lag screw positioning and distal targeting. ADAPT is the only augmented reality instrumentation of its kind.

From March 1, 2021 it becomes mandatory for all orthopedic surgeons at the department to use the ADAPT system when operating pertrochanteric fractures with a gamma3 nail. Following surgery the operating surgeon will fill out the System Usability Scale questionaire and an additional 3 questions.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons who operated patients with pertrochanteric fractures with the use of a gamma3 nail

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons who operated patients with pertrochanteric fractures with the use of a gamma3 nail
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | Questionaire including the "system usability scale" will be send to surgeons within 24 hours following surgery
  Result of the "System Usability Scale" questionaire. The "System Usability Scale" is a questionaire that include 10 questions that participans rank from 1 to 5 (5 means they agree completely, 1 that they disagreee). Highest score is 100 due to the calculation process. Above 80.3 means that the participans are finding ADAPT very usefull and will recommend the use of the system to collegeaus, Above 68 means that participans finds ADAPT usefull, Below 51 means participans finds ADAPT unusefull.

CONTACTS AND LOCATIONS:
Overall Officials: per h gundtoft, md, Principal Investigator — Aarhus University Hospital, orthopedic department
Locations (1):
- Orthopedic Department, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data